CLINICAL TRIAL: NCT07247578
Title: The Link Between Nutrition Education, Behavior, and Body Composition of Women Following a Mediterranean Diet: A Sustainable Approach
Brief Title: The Connection Between Nutrition Education, Behavior, and Body Composition in Women Following a Mediterranean Diet
Acronym: diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ayşe Nur Kahve (Other)
Responsible Party: Sponsor-Investigator, Ayşe Nur Kahve, Lecturer Dr., Aksaray University
Organization: Aksaray University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ANKahve
Record Dates: First submitted 2025-11-15; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Obesity; Sustainability; Education
Keywords: Obesity, Mediterranean diet, sustainability
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Food Choices: Definition of greenhouse gases, Environmentally friendly foods, Environmental impacts of food groups, Definition of water footprint and carbon footprint Reducing Food Waste: Definition of ecological footprint, Definition of food waste, Environmental impacts of food waste, Methods for utilizing food without wasting it, The most wasted foods in the world and Turkey, Ways to reduce food waste Seasonal and local nutrition: Definition of traditional/local foods, The effects of seasonal eating on the human body and the environment The effects of global warming on the environment Purchasing Food: Definition of ecological labels, Definition of expiration dates and recommended consumption dates, The effects of food choices on the environment and the human body
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group receiving sustainable nutrition training (Active Comparator): group receiving sustainable nutrition training
  Interventions: Other: group receiving sustainable nutrition training
- control group (Active Comparator): The group that has not received sustainable nutrition training will be given training at the end of the study.
  Interventions: Other: the group that did not receive sustainable nutrition education

INTERVENTIONS:
Other: group receiving sustainable nutrition training — Sustainable Nutrition Training; Within the scope of this study, face-to-face sustainable nutrition training will be given individually to the trained group by an expert dietitian for 1 hour, once every 2 weeks.
  As part of this study, the group will receive one-hour, face-to-face, individual sustainable nutrition training from a registered dietitian every two weeks. The training flow chart is shown below. Week 1 Educational Topic: Food Choices,Definition of Greenhouse Gases, Environmentally Sensitive Foods, Environmental Impacts of Food Groups, Definition of Water Footprint and Carbon Footprint Week 2 Educational Topic: Reducing Food Waste, Definition of the Ecological Footprint, Definition of Food Waste, Environmental Impacts of Food Waste, Methods for Utilizing Food Without Wasting, The Most Wasted Foods in the World and in Turkey, Ways to Reduce Food Waste Week 3 Educational Topic: Seasonal and Local Nutrition, Definition of Traditional/Regional Foods
  Arms: group receiving sustainable nutrition training
Other: the group that did not receive sustainable nutrition education — The group that has not received sustainable nutrition training will be given training at the end of the study.
  Arms: control group

SUMMARY:
This study aimed to evaluate the effects of Mediterranean Diet and Sustainable Nutrition Education on anthropometric measurements (Weight (kg), BMI, body fat percentage (%), body fat mass (kg), fat-free mass (kg), muscle mass (kg), total body fluid (kg), visceral fat, waist circumference (cm), waist-to-height ratio, and waist-to-hip ratio). It is believed that this education will help bring body composition closer to optimal reference values. This study is expected to reduce energy intake, increase dietary fiber intake, reduce protein from animal sources and increase plant proteins in women's diets, and thus replace saturated fats with monounsaturated fatty acids (MUFAs). This is expected to result in a decrease in body weight and body fat mass.

DETAILED DESCRIPTION:
The Mediterranean diet, in its oldest known definition, is considered a health-promoting dietary model due to its unique characteristics, including regular consumption of unsaturated fats, low-glycemic carbohydrates, high amounts of fiber, vitamins, and moderate amounts of animal-sourced protein. The Mediterranean diet pyramid recommends consuming fish and seafood at least twice a week, 2 servings of white meat, 2-4 servings of eggs, less than 2 servings of red meat, 1 serving or less of processed meat, and less than 3 servings of sweets. Daily, it recommends 2 servings of dairy products, 1-2 servings of seeds and nuts, and increased consumption of spices, herbs, garlic, and onions. It also emphasizes that each main meal should include 1-2 servings of fruit, more than 2 servings of vegetables, olive oil, and 1-2 servings of whole grains. Today, the Healthy Mediterranean Dietary Pattern is included in the 2020-2025 version of the Dietary Guidelines for Americans, not only in the Mediterranean region where its name originates, but also because it is considered a variation of the Healthy American Dietary Pattern. Furthermore, the Mediterranean diet was inscribed on the Representative List of the Intangible Cultural Heritage of Humanity in 2013.

Sustainable diets are diets that preserve and respect biodiversity and ecosystems; are culturally acceptable, accessible, economically feasible and affordable; are nutritionally adequate, safe, and healthy; and make optimal use of natural and human resources. The concept of sustainable food consumption is receiving increasing attention due to global population growth and the threats of climate change. Food production and consumption are among the primary drivers of environmental degradation.

Today, nutritionists emphasize the need to focus on the impact of nutrition on human health, the environment, and food, in contrast to dietary guidelines. Studies examining sustainable dietary behaviors have increased in recent years. Several mechanisms may explain the link between healthier and more sustainable dietary choices and education. Education can be conducive to sustainable diets (e.g., reducing meat consumption) because it encourages the ability to seek and utilize new sources of information, including nutritional information.

In recent years, there has been a focus on the Mediterranean diet's suitability as a sustainable nutrition model due to its high content of plant-based foods and its low ecological, carbon, and water footprint.

This planned study sampled women who follow the Mediterranean diet. The aim was to assess their sustainable nutrition behaviors through sustainable nutrition education sessions. Thus, it is unique in that it is the first study in Turkey to evaluate the suitability of the Mediterranean diet as a sustainable nutrition model and to examine women's anthropometric measurements.

ELIGIBILITY:
Inclusion Criteria:

* o Being a woman between 20 and 49 years of age

  * Having a BMI between 25 kg/m2 and 35 kg/m2
  * Not having any conditions that would impair reality testing ability or cognitive functions and prevent interviews or filling out scales
  * Being literate
  * Having agreed to participate in the study and signed the informed consent form.

Exclusion Criteria:

* o Pregnant and breastfeeding women

  * Those who were unable to attend one or more interview sessions
  * Individuals with implanted pacemakers or defibrillators due to the theoretical possibility of interference with device activity due to the current field caused by impedance measurements
  * Those with any chronic disease and diet
  * Those who regularly use medications that affect metabolism
  * Those using insulin and oral antidiabetic medications
  * Those with allergies or intolerances to any food components of the Mediterranean diet (walnuts, hazelnuts, peanuts, almonds, etc.)
  * Those with a psychiatric illness diagnosed by a physician.

Ages: 20 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Body mass index | 8 weeks
  Body mass index (BMI) will be calculated by dividing body weight by height in square meters and will be evaluated according to the WHO classification for adults.

SECONDARY OUTCOMES:
Body fat percentage | 8 weeks
  Individuals body weight and body composition will be measured using foot-to-foot bioelectrical impedance analysis (BIA). Body fat percentage (% fat) will be measured using the TANITA MC 580.
body fat mass | 8 weeks
  Individuals body weight and body composition will be measured using foot-to-foot bioelectrical impedance analysis (BIA).Body fat mass will be measured using the TANITA MC 580.
visceral adiposity | 8 weeks
  Individuals body weight and body composition will be measured using foot-to-foot bioelectrical impedance analysis (BIA). Visceral adiposity, will be measured using the TANITA MC 580.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe N Kahve, lecturer, Principal Investigator — Aksaray University
Locations (1):
- Eda Ocak Nutrition and Diet Consultancy, Konya, Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF
Time Frame: June 2025-September 2025
Access Criteria: Working at a recognized academic institution, university, research hospital or public research organization.

REFERENCES:
- See also: R Core Team. (2021). R: A language and environment for statistical computing. R Foundation for Statistical Computing, Vienna, Austria. — http://www.R-project.org